CLINICAL TRIAL: NCT04376970
Title: Treatment of Subepithelial Infiltrates Secondary to Epidemic Keratoconjunctivitis: Corticosteroids Versus Cyclosporine Eyedrops: A Randomized Double-blind Study
Brief Title: Treatment of Corneal Infiltrates Secondary to Epidemic Keratoconjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Military Hospital of Tunis (Other)
Responsible Party: Principal Investigator, Asma Khallouli, Teaching hospital assistant lecturer in ophthalmology and a member in the research committee of the military hospital of Tunis, Military Hospital of Tunis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UR17DN02
Record Dates: First submitted 2020-05-02; First posted 2020-05-06 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Adenoviral Keratoconjunctivitis
Keywords: adenoviral keratoconjunctivitis; corticosteroid; cyclosporine; cornea; subepithelial infiltrates
MeSH Terms: conditions — Corneal Diseases | interventions — Fluorometholone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The allocation sequence of the treatment was generated by chance and concealed until all the study was over and all outcomes were assessed. Consecutive patients with subepithelial infiltrates were randomly allocated to one of the two groups by a parallel assignment (1:1).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fluorometholone group (Active Comparator): This group included 38 patients treated with topical fluorometholone 0.1% (FLUCON®) 4 times a day for one month then 3 times a day for one month and 2 times a day for four months.
  Interventions: Drug: FLUCON®
- Cyclosporine A group (Active Comparator): This group included 34 patients treated with cyclosporine A 0.5% eye drops prepared in Ricin oil by the pharmacy of Tunis Military Hospital and prescribed 4 times a day for one month then 3 times a day for one month and 2 times a day for four months.
  Interventions: Drug: Cyclosporine A eye drops 0.5%

INTERVENTIONS:
Drug: FLUCON® — The drug was prescribed monthly according to the predefined regimen. It was not namely specefied in the prescription and was delivered by the hospital pharmacy according to the randomisation list.The subjects were masked to the contents and were instructed to return the empty tubes on monthly visit, wherein 1 pack of topical treatment was provided to them. Neither the patient nor the ophthalmologist knew the allocated treatment. No other medication was allowed during the trial. Duration of the whole regimen was six months. The study included an extra month after the end of the regimen. It was called " wash-out ". Patients who had less than one month of treatment or an uncontrolled treatment side effect or who presented a degenerative iron line were excluded from the rest of the regimen.
  Other Names: Fluorometholone
  Arms: Fluorometholone group
Drug: Cyclosporine A eye drops 0.5% — The same regimen was prescribed for both treatments in order to preserve the double-blind characteristic. Cyclosporine eye drops 0.5%, was prepared from an oral solution of cyclosporine (Sandimmun®) and combined with castor oil, both sterilized by filtration. The preparation was carried out in a pharmacotechnical laboratory where a controlled atmosphere area was dedicated to ophthalmic preparations. The castor oil-Sandimmun® solution mixture is made in a sterile receptacle. After stirring, the mixture is distributed into sterile low density polyethylene bottles. A sterile insert and cap including a tamper-evident seal were placed on each bottle. A content control was then carried out on each batch produced. A sterility test was done on a batch of each day of preparation. Each bottle of each batch is then cleaned, polished, labeled and then packaged in a pre-printed box with an adapted notice. The stability was fixed at 6 months before opening and at 15 days after opening.
  Other Names: CsA
  Arms: Cyclosporine A group

SUMMARY:
Purpose:

To compare efficiency and tolerance between topical 0.5% cyclosporine A and fluorometholone in patients with subepithelial corneal infiltrates (SEIs).

Methods :

A prospective double-blind randomized study was conducted involving 72 eyes, 38 treated with topical fluorometholone and 34 eyes treated with cyclosporine A 0.5% eyedrops, having SEIs. Treatment was considered successful if there was reduction of SEIs and improvement in visual acuity (two snellen lines). Tolerance was mainly evaluated by Schirmer test, conjunctival hyperemia and burning sensation upon eyedrops instillation.

DETAILED DESCRIPTION:
This study was performed on the 72 eyes of 51 patients who were referred to our clinics for epidemic keratoconjunctivitis (EKC).Diagnosis of EKC was based on the constellation of clinical features. The investigators conducted a double-blind randomized prospective parallel trial involving : 38 patients treated with topical fluorometholone and 34 eyes treated with cyclosporine A 0.5% eye drops. Cyclosporine A eye drops were prepared in Ricin oil by the pharmacy of Tunis Military Hospital. The sample size was measured by our research department, to obtain a conclusion of non-inferiority of cyclosporine A compared to fluorometholone in the chronic phase of EKC.

Duration of the whole regimen was six months. The study included an extra month after the end of the regimen. It was called " wash-out ". Patients who had less than one month of treatment or an uncontrolled treatment side effect or who presented a degenerative iron line were excluded from the rest of the regimen.The regimen was the same for both treatments in order to preserve the double-blind characteristic : 4 times a day for one month then 3 times a day for one month and 2 times a day for four months.

Patients were examined on admission to the study and one month , three months, six months and seven months after the onset of treatment. The investigators followed a double-masked fashion in all the phases of the study.

Information gathered in M0 included basic demographic information (age and sex), medical and ophtalmological history, involved eye(s) and duration of symptoms in the acute episode. The investigators evaluated and recorded the interval of time between the onset of the infection and the beginning of the trial and called it " pretherapeutic period ". At each visit, SEIs were photo-documented, best corrected visual acuity (converted to mean logarithm of the minimum angle of resolution), spheric equivalent, SEIs number, intraocular pressure (with non contact tonometers), break-up time and Schimer test type 1 and cup/disc score were recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients having subepithelial infiltrates following epidemic keratoconjunctivites persisting for 14 days or more

Exclusion Criteria:

* a past history of glaucoma or other anterior or posterior segment disease or surgery
* a chronic use of topical or systemic medications
* pregnancy,
* contact lens wearers,
* patients who couldn't attend at least two regimen visits

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in subepithelial infiltrates number | day 0, Month 1, Month 3, Month 6, Month 7
  The subepithelial infiltrates were counted at baseline and at each control visit.The mean change was then calculated between each two visits. Treatment was considrerd efficient if the subepithelial infiltrates decreased half the baseline number or completely disappeared.
Mean change from baseline in Schirmer type 1 value | day 0, Month 1, Month 3, Month 6, Month 7
  The Schirmer value was assessed without local anesthesia. Treatment was considered efficient with a good tolerance when the schirmer type 1 was superior than 5ml/5min.

SECONDARY OUTCOMES:
Mean change from baseline in best corrected visual acuity | day 0, Month 1, Month 3, Month 6
  A gain of two snellen lines from baseline was considered a mark of treatment efficiency.
Mean change from baseline in spheric equivalent | day 0, Month 6
  Spheric equivalent was calculated using an automatic refraction. An increase from baseline of 0.25 dioptries was considered a mark of treatment efficiency.
Mean change from baseline in clinical score | day 0, Month 1, Month 3, Month 6
  These subjective variables : (1) photophobia; (2) Foreign body sensation ; (3) Visual blurring ; (4) tearing and (5) ocular pain were evaluated according to their severity (0 indicated no ; 1, mild ; and 2, severe). The sum of these variables was calculated for each visit and called clinical score.
Overall satisfaction with treatment subjective evaluation: scale | Month 7
  For subjective evaluation of the treatment, patients were asked to evaluate in the seventh month their overall satisfaction with treatment on a scale of 0-10. 0 means no satisfaction with the treatment and 10 means an excellent satisfaction with the treatment.
Number of participants with burning sensation upon eyedrops instillation | day 0, Month 1, Month 3, Month 6
  Burning sensation upon eyedrops instillation was considered as a treatment intolerance mark.
Mean change from baseline in intraocular pressure | day 0, Month 1, Month 3, Month 6
  Intraocular pressure was measured with with non contact tonometers. An increase of 6 mmHg from baseline value was defined as a steroid-induced glaucoma.
Number of participants with appearance of lens opacification and corneal ulcer or superinfection | up to six months
  Lens opacification and corneal ulcer or superinfection were considered as a mark of corticosteroid intolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Afef Maalej, Study Director — Military Hospital of Tunis
Locations (1):
- Military Hospital of Tunis, Tunis, Illinois, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levinger E, Slomovic A, Sansanayudh W, Bahar I, Slomovic AR. Topical treatment with 1% cyclosporine for subepithelial infiltrates secondary to adenoviral keratoconjunctivitis. Cornea. 2010 Jun;29(6):638-40. doi: 10.1097/ICO.0b013e3181c33034. PMID 20458220
- [Result] Maychuk DY, Vasil'eva OA, Russu LI, Mezentseva MV. [Clinical and immunological comparisons of therapeutic regimens for corneal infiltrates secondary to adenoviral keratoconjunctivitis]. Vestn Oftalmol. 2015 Jul-Aug;131(4):49-55. doi: 10.17116/oftalma2015131449-55. Russian. PMID 26489119
- [Result] Reinhard T, Godehardt E, Pfahl HG, Sundmacher R. [Local cyclosporin A in nummuli after keratoconjunctivitis epidemica. A pilot study]. Ophthalmologe. 2000 Nov;97(11):764-8. doi: 10.1007/s003470070025. German. PMID 11130165
- [Result] Aydin Kurna S, Altun A, Oflaz A, Karatay Arsan A. Evaluation of the impact of persistent subepithelial corneal infiltrations on the visual performance and corneal optical quality after epidemic keratoconjunctivitis. Acta Ophthalmol. 2015 Jun;93(4):377-82. doi: 10.1111/aos.12496. Epub 2014 Jul 6. PMID 25043311
- [Derived] Gouider D, Khallouli A, Maalej A, Yousfi MA, Ksiaa I, Bouguerra C, Ajili F, Khairallah M. Corticosteroids Versus Cyclosporine for Subepithelial Infiltrates Secondary to Epidemic Keratoconjunctivitis: A Prospective Randomized Double-Blind Study. Cornea. 2021 Jun 1;40(6):726-732. doi: 10.1097/ICO.0000000000002589. PMID 33201059